CLINICAL TRIAL: NCT04333784
Title: The Effect of Blood Flow Restriction Training on Muscle Thickness and Symptoms in Patients With Rotator Cuff Tendinopathy
Brief Title: Blood Flow Restriction Training in Patients With Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Kara, PhD candidate, Research assistant, Hacettepe University
Other Study IDs: 2020/02-28 (KA-19146)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Rotator Cuff Tendinosis
Keywords: blood flow restriction training; shoulder pain; rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain | interventions — Exercise; Blood Flow Restriction Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exercise with BFR: Patients with rotator cuff tendinopathy will perform the exercises with a pneumatic cuff and blood flow restricted.
  Interventions: Other: Exercise training
- Control: Patients with rotator cuff tendinopathy will perform the exercises without a pneumatic cuff.

INTERVENTIONS:
Other: Exercise training — Exercise with blood flow restriction (with a pneumatic cuff).
  Other Names: Blood flow restriction training
  Groups: exercise with BFR

SUMMARY:
This study was planned to investigate the effect of blood flow restriction exercise training on shoulder muscle strength and muscle thickness, and to determine the change in pain and symptoms in patients with rotator cuff tendinopathy. Patients in the study group will perform the rehabilitation exercises with a pneumatic cuff and blood flow restricted. The patients in the control group will perform the same exercise program without restricting blood flow.

DETAILED DESCRIPTION:
In recent years, one of the popular applications used for muscle hypertrophy and strength training is low-intensity exercise training called Blood Flow Restriction Training. This exercise training has been shown to allow the benefits of high-intensity training at a much lower intensity. Given the light-load nature and strengthening capacity of this training, it can provide an effective clinical rehabilitation stimulus without the high levels of joint stress. It is suggested that it will be a useful exercise alternative especially in individuals who cannot tolerate high-intensity exercise. Especially patients with shoulder pain cannot tolerate high-intensity exercises in early rehabilitation.

This study was planned to investigate the effect of blood flow restriction exercise training on shoulder muscle strength and muscle thickness, and to determine the change in pain and symptoms in patients with rotator cuff tendinopathy.

Hypothesis 1: There is a difference between exercise training with blood flow restriction and exercise training without blood flow restriction in terms of muscle strength and muscle thickness.

Hypothesis 2: There is a difference between exercise training with blood flow restriction and exercise training without blood flow restriction in terms of shoulder pain and shoulder function.

The study was designed as a randomized-controlled. In order to provide an evenly equal number of individuals and homogeneous gender distribution in the groups blocking and stratification will be used as a randomization method. The sample size was calculated to be an 8% difference in muscle thickness at the end of treatment with 80% power and 5% type 1 error. A total of 26 patients were planned to be included in the study, including 13 volunteers in each group. Patients in the study group will perform the determined exercises with a pneumatic cuff and blood flow restricted. The patients in the control group will perform the same exercise program without restricting blood flow. Informed consent will be obtained from all individuals.

Demographic information (age, gender, body mass index, dominant side, affected side, etc.) of all patients will be recorded. Shoulder pain (rest, night and activity- visual analog scale), shoulder range of motions (goniometer), shoulder function (Shoulder Pain and Disability Index-SPADI), shoulder rotator muscle strength (isokinetic dynamometer-Isomed 2000, D&R Ferstl GmbH, Germany) and supraspinatus, infraspinatus, deltoid, biceps, middle trapezius muscle thickness, and acromio-humeral distance (ultrasonography- Logiq P5, General Electrics, USA) will be evaluated before and after 8 weeks of exercise training.

In the first session of treatment, initial assessments and patient education to reduce shoulder pain (avoiding overhead activities and heavy work, appropriate posture, cold-pack application recommendation) will be performed. Exercise training will start in the second session. Individuals in the groups will have 2 sessions per week, 16 sessions of exercise training for 8 weeks. On other days, patients will continue their home exercises recommended by the physiotherapist.

The blood flow restriction training will be applied to patients in the study group, as defined in the literature, by wearing a pneumatic cuff from the most proximal region of the upper limb. Occlusion pressure will be calculated according to the formula for each patient. [Pressure = 0.4 x (systolic blood pressure) + 2.7 x (shoulder circumference) + 62]. Blood flow restriction training will be performed at 30-40% of the arterial occlusion pressure for the upper limb and total duration of 15 minutes. The amount of occlusion pressure will be re-evaluated every two weeks.

Statistical analyses will perform using SPSS program. Descriptive statistics will be presented with means and standard deviations for numerical data and with numbers (n) and percentages (%) for non-numerical data. The suitability of the data obtained from the patients to the normal distribution will be evaluated by the Kolmogorov-Smirnov test. In the case of the normal distribution of data, comparisons between groups will be tested using repeated-measures analysis of variance (two-way ANOVA). When the parametric test conditions are not met, before-after differences within the group will be calculated and the Mann Whitney U test will be used in the analysis of the differences between the groups. Wilcoxon test will be used in intra-group comparisons before and after treatment. In all analyzes, the significance value will be determined as p=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Being 18-45 years
* Unilateral rotator cuff related shoulder pain
* No symptoms in the contralateral shoulder

Exclusion Criteria:

* Diagnosis of hypertension, cardiovascular diseases, peripheral vascular diseases, deep vein thrombosis history, neurological diseases, systemic inflammation, obesity, diabetes
* Subject has cancer
* Pregnancy status
* Cervical symptoms
* Shoulder range of motion limitation
* Injection to the shoulder joint in the last 6 months
* Individuals who do not agree to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with rotator cuff related shoulder pain (tendinopathy findings in ultrasonographic evaluation).
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Changes in shoulder muscle thickness and acromio-humeral distance | baseline and 8 weeks
  Ultrasonography measurement: supraspinatus, infraspinatus, deltoid, biceps, middle trapezius muscle thickness and acromio-humeral distance.
Changes in shoulder muscle strength | baseline and 8 weeks
  Isokinetic assesment: shoulder rotator muscle concentric strength at 60 º/sec and 180 º/sec speeds.

SECONDARY OUTCOMES:
Changes in shoulder pain: visual analogue scale | baseline and 8 weeks
  Self reported pain at rest, activity and night with 10cm visual analogue scale. 0=no pain, 10=pain as bad as can be.
Changes in shoulder function | baseline and 8 weeks
  Shoulder pain and disability index. It consist of two subscales (pain and disability) are averaged to produce a total score ranging from 0 (best) to 100 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Levent Ozcakar, PhD,Prof., Principal Investigator — Hacettepe University; Irem Duzgun, PhD,Prof., Principal Investigator — Hacettepe University; Dilara Kara, MSc., Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewis J. Rotator cuff related shoulder pain: Assessment, management and uncertainties. Man Ther. 2016 Jun;23:57-68. doi: 10.1016/j.math.2016.03.009. Epub 2016 Mar 26. PMID 27083390
- [Background] Benitez-Martinez JC, Casana-Granell J, de Llago YE, Villaron-Casales C, Espi-Lopez GV, Jimenez-Diaz F. Cross Sectional Area of the Supraspinatus Muscle and Acromio-humeral Distance in Overhead Athletes With and Without Shoulder Pain: A Cross-sectional Study. J Sport Rehabil. 2017 Nov;26(6):524-529. doi: 10.1123/jsr.2016-0146. Epub 2016 Nov 11. PMID 27834581
- [Background] Littlewood C, Malliaras P, Chance-Larsen K. Therapeutic exercise for rotator cuff tendinopathy: a systematic review of contextual factors and prescription parameters. Int J Rehabil Res. 2015 Jun;38(2):95-106. doi: 10.1097/MRR.0000000000000113. PMID 25715230
- [Background] Seitz AL, Podlecki LA, Melton ER, Uhl TL. NEUROMUSCULAR ADAPTIONS FOLLOWING A DAILY STRENGTHENING EXERCISE IN INDIVIDUALS WITH ROTATOR CUFF RELATED SHOULDER PAIN: A PILOT CASE-CONTROL STUDY. Int J Sports Phys Ther. 2019 Feb;14(1):74-87. PMID 30746294
- [Background] Dankel SJ, Jessee MB, Abe T, Loenneke JP. The Effects of Blood Flow Restriction on Upper-Body Musculature Located Distal and Proximal to Applied Pressure. Sports Med. 2016 Jan;46(1):23-33. doi: 10.1007/s40279-015-0407-7. PMID 26446893
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Ladlow P, Coppack RJ, Dharm-Datta S, Conway D, Sellon E, Patterson SD, Bennett AN. Low-Load Resistance Training With Blood Flow Restriction Improves Clinical Outcomes in Musculoskeletal Rehabilitation: A Single-Blind Randomized Controlled Trial. Front Physiol. 2018 Sep 10;9:1269. doi: 10.3389/fphys.2018.01269. eCollection 2018. PMID 30246795
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Background] Thiebaud RS, Loenneke JP, Fahs CA, Rossow LM, Kim D, Abe T, Anderson MA, Young KC, Bemben DA, Bemben MG. The effects of elastic band resistance training combined with blood flow restriction on strength, total bone-free lean body mass and muscle thickness in postmenopausal women. Clin Physiol Funct Imaging. 2013 Sep;33(5):344-52. doi: 10.1111/cpf.12033. Epub 2013 Apr 3. PMID 23701116
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Proximal, Distal, and Contralateral Effects of Blood Flow Restriction Training on the Lower Extremities: A Randomized Controlled Trial. Sports Health. 2019 Mar/Apr;11(2):149-156. doi: 10.1177/1941738118821929. Epub 2019 Jan 14. PMID 30638439
- [Background] Yasuda T, Fujita S, Ogasawara R, Sato Y, Abe T. Effects of low-intensity bench press training with restricted arm muscle blood flow on chest muscle hypertrophy: a pilot study. Clin Physiol Funct Imaging. 2010 Sep;30(5):338-343. doi: 10.1111/j.1475-097X.2010.00949.x. Epub 2010 Jul 4. PMID 20618358
- [Background] Van Roekel HE, Thurston AJ. Tourniquet pressure: the effect of limb circumference and systolic blood pressure. J Hand Surg Br. 1985 Jun;10(2):142-4. doi: 10.1016/0266-7681(85)90002-6. PMID 4031590
- [Background] Land H, Gordon S, Watt K. Isokinetic clinical assessment of rotator cuff strength in subacromial shoulder impingement. Musculoskelet Sci Pract. 2017 Feb;27:32-39. doi: 10.1016/j.msksp.2016.11.012. Epub 2016 Dec 10. PMID 28637599
- [Derived] Kara D, Ozcakar L, Demirci S, Huri G, Duzgun I. Blood Flow Restriction Training in Patients With Rotator Cuff Tendinopathy: A Randomized, Assessor-Blinded, Controlled Trial. Clin J Sport Med. 2024 Jan 1;34(1):10-16. doi: 10.1097/JSM.0000000000001191. Epub 2023 Sep 14. PMID 37706671